CLINICAL TRIAL: NCT07327827
Title: Effects of Back School Based Intervention Versus Cranio-Cervical Muscle Training on Pain, Posture and Disability in Computer Users With Cervicogenic Headache
Brief Title: Comparative Effects of Back School Based Intervention Versus Cranio-Cervical Muscle Training in Computer Users With Cervicogenic Headache
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Principal Investigator, Dr. Hufsa Tariq, Assistant Professor, Lahore University of Biological and Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UBAS/ERB/FoRS/25/029
Record Dates: First submitted 2025-12-25; First posted 2026-01-08 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Cervicogenic Headache
Keywords: Cervicogenic Headache; Back School Based Program; Cranio-Cervical Muscle Training; Pain; Posture; Headache; Disability
MeSH Terms: conditions — Post-Traumatic Headache; Pain; Headache

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Back School Based Intervention (Experimental): Back School Based Intervention
  Interventions: Other: Back School Based Intervention
- Cranio- Cervical Muscle Training (Active Comparator): Cranio- cervical muscle Training
  Interventions: Other: Cranio-Cervical muscle Training

INTERVENTIONS:
Other: Back School Based Intervention — * Patient will receive 2 sessions per week for 8 weeks for a total of 16 sessions. Each session lasted for 35 minutes.
  * Conventional Physical therapy will be provided in which stretching of the tight muscles which include SCM, upper trapezius, levator scapulae, scalene, sub occipitals, pectoralis minor, and pectoralis major. Neck stretches, chin tucks, scapular squeezes, and upper back strengthening exercises with 5 repetitions will be performed. Trigger points of sub occipitals, SCM, and temporalis are released because they cause headache.
  * Back School Based Intervention includes both theoretical and practical part. Patients had total of 16 sessions out of which 14 will be practical one and remaining two will be theoretical one. In theoretical part main focus is on the patient education and guidance. In practical part resistive exercises of increase intensity in each session will be performed in which main focus is on the strengthening
  Arms: Back School Based Intervention
Other: Cranio-Cervical muscle Training — * Patient will receive 2 sessions per week for 8 weeks for a total of 16 sessions. Each session lasted for 35 minutes. Conventional physical therapy will be same in both groups
  * Cranio- cervical muscle training session main focus is on the strengthening and posture correction. Cervical flexion, extension and stabilization exercises will be performed which helps to strength muscles and helps to neutralize posture and ultimately disability which is due to headache will be reduced.
  Arms: Cranio- Cervical Muscle Training

SUMMARY:
The aim of the study is to compare Back School Based Intervention with Cranio- Cervical muscle training in participants with Cervicogenic headache. The study wants to investigate that which intervention helps to mange pain, improve posture and reduce disability. The study aims to answer the question:

* How effective is Back School Based intervention on pain, posture and disability in computer users with Cervicogenic headache compared to Cranio-cervical Muscle Training? Participants will
* Attend the treatment sessions of the group in which they are placed.
* Take treatment session two times a week for eight weeks.
* Participants will be asked about their pain and activities throughout the study.

DETAILED DESCRIPTION:
* Headache is one of the disorder that affects 50% of the population worldwide which have negative impact on the quality of life. Cervicogenic headache is the secondary type of headache in which the pain referred from the cervical spine. Headache aggravates by the neck movement and significant reduced range of motion is noticed among patients.
* The management of the cervicogenic headache is both pharmacological and non- pharmacological but pharmacological having more side effects.Non pharmacological management includes massage, dry needing, physical therapy exercises, manual therapy and patient education.
* Cranio-cervical muscle training include cranio-cervical flexion exercises, strengthening, stretching, posture exercises and cervical stabilization exercises. These exercises altogether helps in the strengthening of the neck and shoulder muscles which ultimately correct the cervical impairment which neutralize the posture and decrease the load on the structures of the spine.
* Back school based exercise program can have both practical and theoretical sessions. In practical part patient is guided to the different strengthening and flexibility exercises with increase resistance in each session. In theoretical part patient education is the main part. Patient is educated about the anatomical and posture related changes in the spine so he/ she can identify and correct them by incorporating in their daily life.

ELIGIBILITY:
Inclusion Criteria:

* Participants of both gender.
* Participants aged between 19 to 44 years.
* Participants having unilateral headache without side shift for>3 months aggravated by neck movement.
* Participants with pain intensity ≥3 on a visual analog scale (VAS).
* Participants working on the computer for an average 32 h per week.
* Participants having positive cervical flexion rotation test (CFRT).
* Participants having joint tenderness in at least one of the upper three cervical joints with palpation.

Exclusion Criteria:

* If participants having any history of fractures or previous surgery of the vertebral column, any degenerative and inflammatory arthritis, osteoporosis, dislocations, cervical radiculopathy/myelopathy and any history of whiplash injury.
* Participants showing any signs of the five 'D's' or three 'N's.

Ages: 19 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-01-23 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-07-18 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue scale | It will be measured at baselines, 4 weeks and at 8 weeks.
  Visual Analogue Scale is used for the measurement of pain.a hand written mark on 10 cm line helps to differentiate pain in different patients. If Patient reports minimum pain level more than 3 than considered as the patient required for study maximum pain level will be 10
Headache Disability Index | It will be measured at baseline, 4 weeks and at 8 weeks.
  Headache Disability Index is used to evaluate the impact of headache on person's daily life activities. It consists of 25 questions. Patient answer the question as yes scored as 4, sometimes as 2 or no as 0. The score interpretation for disability is measured and for mild disability it is 10 to 28, for moderate disability is 30 to 48, for severe disability is 50 to 68 and for complete disability 72 or higher is noticed.
Plumb Line Assessment of Posture | It will be measured at baseline, 4 weeks and at 8 weeks.
  A plumb line is used as reference to measure the abnormality or deviation from posture. It helps to pinpoint those areas of the body which are away from neutral alignment of the body such as rounded shoulder, forward head posture and abnormal tilt of pelvis. Patient reported as deviated or non deviated from neutral posture.
Cervical Flexion Rotation Test | It will be measured at baseline, 4 weeks and at 8 weeks.
  Cervical flexion rotation test is used to determine the presence of joint dysfunction at the C 1/2 level. The cervical spine is fully flexed to avoid rotational movements then rotated to right and left to find out any pain or restrictions in the joints. Pain provocation and limited rotation indicate the positive test result. Maximum range of rotation will be 45 which is considered as normal. Range less than 45 will need to be corrected.

CONTACTS AND LOCATIONS:
Overall Officials: Laiba Azam, Principal Investigator — Lahore University of Biological and Applied Sciences
Locations (1):
- Sir Ganga Ram Hospital Lahore, Lahore, Punjab Province, Pakistan